CLINICAL TRIAL: NCT04730661
Title: Efficacy of the Sit to Stand Test (STST) in the Decision to Hospitalize a Patient Consulting the Emergency Department for COVID 19 (Coronavirus Infectious Disease)
Brief Title: Efficacy of the Sit to Stand Test in the Decision to Hospitalize a Patient Consulting the Emergency Dept for COVID 19
Acronym: SITCOV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decrease of inclusion capacities because of the control of COVID 19 epidemia thanks to vaccination
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020/0339/HP
Record Dates: First submitted 2021-01-19; First posted 2021-01-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm (No Intervention): For the patients enrolled in this conventional arm, the decision of hospitalisation or discharge will be taken with usual criteria (pulsed oxygen saturation (SpO2) in room air <92% and respiratory rate> 22/min, respiratory rate> 30/min, Blood gas hypoxemia, decompensation of comorbidity, home monitoring not possible, other intercurrent pathology requiring hospitalization, several risk factors for COVID infection requiring hospitalization in intensive care (age> 65y, hypertension complicated by a cardiovascular event, chronic cardiovascular disease, unbalanced diabetes with complications, chronic respiratory disease (excluding well-controlled asthma), chronic renal failure dialysis, obesity, progressive cancer under treatment, congenital or acquired immunosuppression)
- Interventional arm (Experimental): For the patients enrolled in this interventional arm, the decision of hospitalisation or discharge will be taken with usual criteria and the result of Sit to Stand Test.
  Interventions: Diagnostic Test: Sit to stand test

INTERVENTIONS:
Diagnostic Test: Sit to stand test — The sit to stand test (or STST) is a test consisting of performing as many sit-to-stand tests as possible in one minute, from a chair without armrests.
  We note before and during this test, the SpO2 (pulsed oxygen saturation) (rest value and minimum value during exercise), heart rate (HR), dyspnea on the modified Borg scale as well as the number of chair lifts performed. completely and minimum SpO2 during the recovery phase.
  The possible results from this one-minute test are as follows:
  * If SpO2 <90% or appearance of signs of respiratory distress: Immediate stop of the test and hospitalization
  * SpO2 <90% or decrease in SpO2 ≥ 4% during the test or during the recovery period: Hospitalization
  * SpO2 ≥90% and no decrease in SpO2 ≥ 4% during the test or during the recovery period which will be 3 minutes maximum: discharge.
  Arms: Interventional arm

SUMMARY:
As part of the Coronavirus Infectious Disease 2019 (COVID19) pandemic, the hospital care system is facing a major strain. Patients with SARS-Cov2 (severe acute respiratory syndrome coronavirus 2 ) infection can worsen very quickly, possibly presenting, within hours, severe respiratory failure requiring urgent specialized care. Therefore, it is essential to develop emergency assessment tools to assess relevant criteria to decide which patients must be kept under hospital monitoring and which patients can be treated on outpatient care.

The aim of this study is to assess the efficacy of STST in the decision to hospitalize patients consulting emergency department for a SARS-Cov2 infection. The investigators wish to show that the addition of this test to the usual hospitalization criteria reduces the proportion of patients hospitalized 48 hours after their first visit to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Admit to emergency department for suspected SARS-Cov2 infection
* SARS-CoV2 infection confirmed by Real Time Polymerase Chain Reaction (RT - PCR) before the first discharge of emergency department
* Patient affiliated or beneficiary of a health care insurance
* Effective contraception in women of childbearing age. For postmenopausal women, amenorrhea for at least 12 months before the inclusion visit

Exclusion Criteria:

* Patient presenting criteria for admission to intensive care: signs of acute respiratory distress , respiratory rate> 30 / min, oxygen dependence > 6L / min on face mask for an SpO2 ≥ 95% or an arterial oxygen pressure >8kPa, neurological disorders, systolic blood pressure (SBP) <90mmHg despite fluid resuscitation, lactates> 2mmol / L, bradycardia, or heart rate disorders
* Patient with SpO2 <90% in spontaneous ventilation in room air at rest
* Patient with functional impairment or deterioration of the general condition leading to the inability to perform STST
* Patient with a resting SBP> 180 mmHg or resting diastolic blood pressure (DBP)> 100 mmHg or resting heart rate (HR)> 120 / min
* Patient with decompensated or unbalanced cardiac pathology
* Patient previously included in the study following a previous admission to emergency department
* Patient deprived of liberty, unable to consent freely
* Patient non affiliated or beneficiary of a health care insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Proportion of late hospitalizations, within 48 hours of first discharge from emergency department, and motivated by worsening symptoms secondary to SARS-Cov2 infection. | 7 days

SECONDARY OUTCOMES:
Proportion of immediate hospitalizations after the 1st admission at emergency department. | 7 days
Proportion of adverse events related to SARS-Cov2 infection within 7 days of patient inclusion. | 7 days
  The adverse events identified are:
  * medical consultation,
  * readmission to the emergency department,
  * hospitalization,
  * hospitalization in intensive care unit,
  * death.
Establish the correlation between the number of chair rises performed on STST and the occurrence of an adverse event. | 7 days
  The adverse events identified are:
  * medical consultation,
  * readmission to the emergency department,
  * hospitalization,
  * hospitalization in intensive care unit,
  * death.
Correlation between SpO2 and the occurrence of an adverse event | 7 days
  the difference between the measurement of SpO2 before and after STST will be used to establish the correlation between this difference and the occurrence of an adverse event.
Correlation between heart rate (HR) and the occurrence of an adverse event | 7 days
  the difference between the measurement of HR before and after STST will be used to establish the correlation between this difference and the occurrence of an adverse event.
Correlation between dyspnea score and the occurrence of an adverse event | 7 days
  the difference between the measurement of dyspnea score before and after STST will be used to establish the correlation between this difference and the occurrence of an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARTAUD-MACARI, MD, Principal Investigator — Pneumology, Thoracic Oncology and Respiratory Intensive Care Unit; Fairuz BOUJIBAR, PhD, Study Director — Thoracic Surgery
Locations (1):
- Rouen university hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No